CLINICAL TRIAL: NCT03934086
Title: BHV3000-401: An Open-label, Intermediate-size, Expanded Access Study of BHV-3000 in the Acute Treatment of Migraine
Brief Title: An Open-label, Intermediate Size, Expanded Access Study of BHV-3000 in the Acute Treatment of Migraine
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: BHV3000-401
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Migraine
Keywords: Migraine prevention, phonophobia, photophobia, nausea
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea | interventions — rimegepant sulfate

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: rimegepant — rimegepant 75 mg

SUMMARY:
The purpose of this protocol is to allow subjects who completed any BHV3000 (rimegepant) clinical study to continue to have access to rimegepant while collecting ongoing safety data.

(NOTE: ONLY FOR PATIENTS who participated in a previous BHV-3000/Rimegepant Clinical Trial in the past)

ELIGIBILITY:
Inclusion Criteria:

1.Subjects who have completed any BHV3000 (rimegepant) clinical study without significant protocol violations.

Exclusion Criteria:

1. History of basilar migraine or hemiplegic migraine
2. History with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease
3. HIV history
4. Uncontrolled hypertension or uncontrolled diabetes
5. Current diagnosis of major depression, other pain syndromes, psychiatric conditions (e.g., schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments
6. History of gastric, or small intestinal surgery, or has a disease that causes malabsorption

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult